CLINICAL TRIAL: NCT03869138
Title: Alternative Therapies for Improving Physical Function in Individuals With Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Tanvi Bhatt, Assistant Professor, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0035
Record Dates: First submitted 2019-03-01; First posted 2019-03-11 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Masking Description: Intervention provider and assessor were all blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Virtual-reality based dance group (Experimental): Virtual-reality based dance training - Participants received Virtual-reality based dance training for 6 weeks using the commercially available Kinect dance game (Microsoft Inc., Redmond, WA, U.S.A.) "Just Dance 3". The six week session consisted of 5 sessions/week, next two weeks of 3 sessions/week and last two weeks of 2 sessions/week, for a total of 20 sessions. Participants played on 10 songs for the first 2 weeks, progressing to 12 songs during the 3nd and 4th weeks with an addition of 2 more songs of their choice during the last two weeks. Participants played on alternating slow- and fast-paced songs (each maximum of 4 minutes in duration) with a five minutes break after a set of one slow and fast song.
  Interventions: Behavioral: Virtual-reality based dance training

INTERVENTIONS:
Behavioral: Virtual-reality based dance training — Participants will receive therapy using the "Just Dance" using the commercially available Kinect gaming system (Microsoft Inc, Redmond, WA, USA. Each song involves repetitive action for each dance step (at least 20 repetitions over the entire song) and visual cues on the screen (a stick figure at the bottom right) indicating the upcoming dance step. Participant's playing the game to reduce risk of exercise related adverse effects. Participants will dance on 10 songs starting from a slow-pace progressing to a medium pace (each max 5 minutes long). Participants will receive 5 minutes rest after playing on each song. This will be conducted by two physical therapists.
  Other Names: VR-based dance,; exergaming-based dance

SUMMARY:
Neurological impairment is a devastating disease for patients and their families and a leading cause of adult disability. Traditional rehabilitative therapies can help regain motor function and ameliorate disability. However, health care reimbursed rehabilitation is usually provided for up to 6 months post stroke (3 months in form of inpatient therapy and 3 months in outpatient therapy). There are increasing community and other facilities offering rehabilitation in form of conventional, recreational and alternative (Yoga, Tai-chi) therapy. However, implementation of these conventional therapy techniques in individuals with neurological disorder impairments is tedious, resource-intensive, and costly, often requiring transportation of patients to specialized facilities. Based on recent evidence suggesting significant benefits of repetitive, task-orientated training, investigators propose to evaluate the feasibility of an alternative dance and gaming based virtual dance and gaming based therapy to improve overall physical function of community-dwelling individuals with neurological impairments, compared to conventional therapeutic rehabilitation. This pilot study aims to systematically obtain pilot data on compliance and efficacy as well as performing power analysis and sample size calculation for developing it into a randomized controlled trial for extramural funding purposes. The objective of the study is to determine the safety, feasibility, compliance and efficacy of an alternative dance and gaming-based virtual gaming therapy to improve overall physical function of community-dwelling individuals with neurologically impairment and compare it to that of conventional rehabilitation and also to determine the gains in community participation and integration with longer-term compliance to the dance and gaming -based intervention.

DETAILED DESCRIPTION:
This pilot study aims to systematically obtain pilot data on compliance and efficacy as well as performing power analysis and sample size calculation for developing it into a randomized controlled trial for extramural funding purposes. Aim 1: To determine the efficacy of an alternative dance and gaming based cognitive-motor virtual reality therapy to that of a conventional rehabilitation in a clinical setting to improve physical and cognitive function of healthy adults and neurologically impaired community-dwelling individuals under both short duration high intensity and long duration intervention paradigm. The primary safety outcome would be the proportion of patients experiencing intervention-related adverse events during the study period. The primary feasibility outcome would be the total time receiving intervention (i.e. compliance). Motivation index found to correlate highly with compliance will be evaluated by the self-report Intrinsic Motivational Inventory and serve as the secondary factor. The primary efficacy outcome measures to determine improvements in physical function would incorporate main domains: Sensorimotor impairment and function (upper and lower extremity), balance control and fall-risk, cognition, cardiovascular function, and community participation and integration administered pre and post intervention (details in methods). Hypothesis 1: Investigators hypothesize that alternative dance and gaming based cognitive-motor virtual reality therapy and perturbation training would show greater efficacy through improvement in main domains of physical function (sensorimotor, balance control, cognition, fall-risk, and cardiovascular function) compared to the conventional balance training. Aim 2: To determine the compliance and gains in community participation and integration following gaming based virtual reality intervention. Hypothesis 2: With same number of sessions of both types of training, investigators hypothesize that virtual reality based interventions would show better compliance to therapy through better score on Intrinsic Motivational Inventory (IMI) than the conventional therapy. Higher IMI scores in this virtual reality intervention group will be positively correlated with the improvements in quality of life (Motor Activity Log), Community integration (CIQ) and Fall-risk reduction (Falls Efficacy and Activities-specific balance confidence scales).

Aim 3: To compare the compliance and effect of a short duration high intensity training (20 sessions over 6 weeks) with a low intensity longer duration (36 sessions over 12 weeks) balance training for the two types of interventions. Hypothesis 3: It is hypothesized that for both types of interventions, short duration high intensity training will be as effective for improvement in physical function as longer duration low intensity training. However, the compliance of short duration training would be greater (higher IMI score) compared to the longer duration training.

ELIGIBILITY:
Inclusion Criteria:

1. Participants should be 18 to 90 years of age.
2. Able to follow instructions provided in English.
3. History of neurological impairment (Stroke, Parkinson's disease and Multiple Sclerosis) for at least 6 months prior to evaluation (self-report, confirmed by participant's physician).
4. Able to stand and walk with or without assistive device or braces as part of their activities of daily living (self-report).
5. Cognitive skills to actively participate (score of < 26 on Montreal cognitive assessment indicates cognitive impairment) (30).
6. Stroke - a) Upper extremity limb function (score of at least 25 on the Fugyl Myer Upper extremity test and Muscle performance grade on deltoid, pec major and and triceps of > or = 2/5).
7. Parkinson's disease a) - Stable medication use b) stage I or II of the Boher classification of Parkinson's disease c) No sudden fluctuations (on-off phenomenon).
8. Multiple Sclerosis - No Severe disability "Expanded Disability Status Scale" (EDSS scale < or = 4.5).

Exclusion Criteria:

* 1. Significant cognitive or communicative impairment indicated by a score of > 26 on Montreal cognitive assessment indicates cognitive impairment. In neurologically impaired individuals, for cognitive impairment a score of <25 on Mini Mental State Exam Score; for aphasia <71% on Mississippi Aphasia Screening Test and >15 on Geriatric Depression Scale.

  2. Presence of concurrent severe medical illness, including unhealed pressure sores, active or untreated infection, thromboembolic disease, severe contractures, active heterotrophic ossification in the lower extremities, lower limb fractures, known history of peripheral nerve injury in the lower legs, history of cardiovascular or pulmonary complications, or with pacemakers and history of metabolic (endocrine, hepatic) or renal dysfunction, uncontrolled seizures (Self-report).

  3. History of any acute and significant cardiopulmonary, musculoskeletal or systemic diagnosis in the past 6 months or history of a recent major surgery (<6months) or hospitalization (<3months) and on any sedative drugs.

  4. Partcipants unavailable for 12 weeks of participation, 5. Current participation in other treatment (i.e.- Botox) or other research studies during the phase of the study.

  6. Pregnancy. 7. Uncontrolled pain >3/10 on VAS 8. Complains of shortness of breath 9. Uncontrolled hypertension (systolic blood pressure (SBP) > 165 mmHg and/or diastolic blood pressure (DBP) > 110 mmHg during resting) [1,2].

  10. Resting hear rate (HR) > 85% of age-predicted maximal heart rate (HRmax) (HRmax = 220 - age) [3].

  11. Oxygen saturation (measured by pulse oximeter) during resting < 95%. 12. Severe cardiac disease (New York Heart Association classification of II-IV) [1].

  13. Exclusion Criteria for Laboratory Slip test. i. T score of < -2 on the Bone density, measured through via the heel ultrasound machine. It must be noted that the particpants will be explained that they were excluded from the balance test to avoid any injury risk as there is a chance that their bones may be weak. However, they will be told that the ultrasound test does give more false positives (i.e. lower scores indicating weak bones when in fact they are not weak) and that they probably could see their physician for a more conclusive test (such as the full-body bone scan).

ii. Partcipants with > 250 lbs in weight or with a BMI OF >35Kg/m2. It should be noted that the harness system is capable of tolerating up to 300 lbs of weight safely.

iii. Unable to walk a length of 8 meters without cane two times with a rest break in between the two walks, lasting shorter than five minutes.

iv. Unable to stand for at least 5 minutes (to accommodate length of a dance song) as assessed by decrease in blood pressure by 20 mmHg systolic and 10 mmHg diastolic measured by the a research team member.

Please note that the exclusion criteria for the Laboratory Slip test will only exclude participants from taking this test. They will still be part of the study if other inclusion /exclusion criteria are met and will go through the other tests and the intervention protocol.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-09-09 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Postural Stability | Baseline (week 0), Mid-training (2nd week), and Post-training (7th week)
  Postural Stability can be defined by simultaneous control of center of mass position and velocity during slip-like perturbation relative to the rear edge of base of support (rear heel). The position normalized with the individual's foot length, and velocity by square root of gravitational acceleration and individual's body height. Greater values indicate greater stability.
Compliance to therapy (total time spent over the intervention duration) | Baseline (week 0), Mid-training (2nd week), and Post-training (7th week)
  Compliance will be assessed by logs of participation time (total time summed over the intervention duration). This will assess if participants were able to complete and tolerate the intervention. Higher values indicate more compliance.
Change in reaction time with functional arm reach | Baseline (week 0), Mid-training (2nd week), and Post-training (7th week)
  Reaction time was evaluated with electromyography as the time elapsed between the final cue, "Go" (at 4s), and the onset of EMG signal (calculated as ±1 standard deviation from baseline). Electromyographic will be used to monitor muscle activity in both upper extremities for stand arm reaching. The test will take about 30 minutes.

SECONDARY OUTCOMES:
Change in Movement Velocity | Baseline (week 0), Mid-training (2nd week), and Post-training (7th week)
  Degrees of movement per second of a self-initiated movement. Higher values indicate better performance.
Change in physical activity | Baseline (week 0), Mid-training (2nd week), and Post-training (7th week)
  For this purpose, the number of steps taken for up to one week will be measured using a wearable sensor by Tractivity (Huston, Texas). During the initial visit, participant will be given the sensor placed in an ankle band. After initial activity monitoring for one week, participants will be scheduled for the training session. After the training participants post-training one-week physical activity will also be monitored. Higher number of steps, indicate more physical activity.
Change in Berg Balance Scale | Baseline (week 0), Mid-training (2nd week), and Post-training (7th week)
  Assess static and dynamic balance control. It is a 14 item scale. Score for each item ranges from 0-4. Item score are then summed and maximum score of 54 can be obtained. Less than 45 on this scale indicates a greater risk for falling.

CONTACTS AND LOCATIONS:
Overall Officials: Tanvi Bhatt, Study Director — University of Illinois Chicago
Locations (2):
- United States (2):
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Illinois Chicago, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No